CLINICAL TRIAL: NCT04473898
Title: Telerehabilitation After Covid-19: Effectiveness of Respiratory and Aerobic Training
Brief Title: Telerehabilitation After Coronavirus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KTO Karatay University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: KaratayU2
Record Dates: First submitted 2020-07-14; First posted 2020-07-16 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2020-07

CONDITIONS: COVID
Keywords: Covid-19; Telerehabilitation; Respiratory Exercises; Aerobic Exercises
MeSH Terms: conditions — COVID-19 | interventions — Patient Education as Topic; Breathing Exercises

STUDY DESIGN:
Intervention Model Description: It is planned to include 3 groups in the study. The group 1 will be informed about covid-19 and hygiene. Aerobic exercise will be offered to Group 2, aerobic exercise + breathing exercises will be offered to Group 3. The persons to be included in the groups will be determined randomly.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patient Education Group (Sham Comparator): Information training about COViD-19 and its symptoms, hygiene education, family education
  Interventions: Behavioral: Patient Education
- Aerobic Training Group (Experimental): Teaching and regular follow-up of aerobic exercises shown online
  Interventions: Other: Aerobic Exercise Training; Behavioral: Patient Education
- Aerobic + Respiratory Training Group (Experimental): Teaching and regular follow-up of aerobic and respiratory exercises shown online
  Interventions: Other: Aerobic Exercise Training; Behavioral: Patient Education; Other: Respiratory Exercise Training

INTERVENTIONS:
Other: Aerobic Exercise Training — Aerobic exercises using all body muscles and that one can do on their own after being shown online
  Arms: Aerobic + Respiratory Training Group; Aerobic Training Group
Behavioral: Patient Education — Patient education about covid-19 and hygiene education
Other: Respiratory Exercise Training — Respiratory exercises that one can do on their own after being shown online
  Arms: Aerobic + Respiratory Training Group

SUMMARY:
The aim of the study is to investigate the effects of telerehabilitation program on COVID-19 symptoms, quality of life, level of depression, perception of dyspnea, sleep, fatigue, kinesiophobia and patient satisfaction in individuals diagnosed with COVID-19.

DETAILED DESCRIPTION:
Because of the risk of infection, telerehabilitation applications are recommended for patients with COVID-19. There are no studies in the literature evaluating the effectiveness of telerehabilitation program after COVID-19. In particular, the importance of the first eight weeks after the disease was emphasized.

It is thought that the telerehabilitation program will improve the functional capacities and quality of life of patients in order to adapt to the daily life after the infection more easily, to cope with the symptoms brought about by the disease more easily and to prevent the respiratory distress, intensive care stay and inactivity due to muscle weakness.

ELIGIBILITY:
Inclusion Criteria:

* volunteering to participate in the study
* at least once diagnosed with COVID-19,
* has a cognitive level that can adapt to online exercises,
* having a physical condition suitable for exercises
* staying in hospital due to covid-19

Exclusion Criteria:

* refuse to participate in the study
* having neurological, cardiac, respiratory disease that prevents exercise

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2020-06-19 (Actual); Primary Completion 2020-10-19 (Actual); Study Completion 2021-02-17 (Actual)

PRIMARY OUTCOMES:
Dyspnoea | baseline
  It will be evaluated by the Modified Medical Research Council (mMRC). It consists of 5 items between 0 and 4. The increase in the score indicates the severity of dyspnea.
Anxiety and Depression | baseline
  It will be evaluated by the Hospital Anxiety and Depression Scale (HADS). The questionnaire comprises seven questions for anxiety and seven questions for depression, and takes 2-5min to complete. Although the anxiety and depression questions are interspersed within the questionnaire, it is vital that these are scored separately. Cut-off scores are available for quantification, for example a score of 8 or more for anxiety. The increase in the score indicates the severity of anxiety and depression.
Sleep Quality | baseline
  It will be evaluated by pittsburgh sleep quality index
Health Related Quality of Life | baseline
  It will be evaluated by SF-36
Dyspnoea | 6 weeks later
  It will be evaluated by the Modified Medical Research Council (mMRC). It will be evaluated by the Modified Medical Research Council (mMRC). It consists of 5 items between 0 and 4. The increase in the score indicates the severity of dyspnea.
Anxiety and Depression | 6 weeks later
  It will be evaluated by the Hospital Anxiety and Depression Scale (HADS). The questionnaire comprises seven questions for anxiety and seven questions for depression, and takes 2-5min to complete. Although the anxiety and depression questions are interspersed within the questionnaire, it is vital that these are scored separately. Cut-off scores are available for quantification, for example a score of 8 or more for anxiety. The increase in the score indicates the severity of anxiety and depression.
Sleep Quality | 6 weeks later
  It will be evaluated by pittsburgh sleep quality index
Health Related Quality of Life | 6 weeks later
  It will be evaluated by SF-36

SECONDARY OUTCOMES:
Kinesiophobia | baseline
  It will be evaluated by Kinesiophobia Causes Scale. The questionnaire consist of 20 closed questions, assessed in a range from 0 to 100 - a higher score indicating a higher fear of movement
Patient Satisfaction | 6 weeks later
  It will be evaluated by patient satisfaction scale. Likert scale questionnaire proposed seven dimensions of patient satisfaction directed toward their doctors. These are general satisfaction, technical quality, interpersonal manner, communication, financial aspects, time spent with doctor, and accessibility and convenience. Increased score indicates decreased satisfaction. The minimum score is 18, the maximum score is 90.
Fatigue | baseline
  It will be evaluated by Fatigue Severity Scale. A self-report scale of nine items about fatigue, its severity and how it affects certain activities. Answers are scored on a seven point scale where 1 = strongly disagree and 7 = strongly agree. This means the minimum score possible is nine and the highest is 63.
Kinesiophobia | 6 weeks later
  It will be evaluated by Kinesiophobia Causes Scale. The questionnaire consist of 20 closed questions, assessed in a range from 0 to 100 - a higher score indicating a higher fear of movement
Fatigue | 6 weeks later
  It will be evaluated by Fatigue Severity Scale. A self-report scale of nine items about fatigue, its severity and how it affects certain activities. Answers are scored on a seven point scale where 1 = strongly disagree and 7 = strongly agree. This means the minimum score possible is nine and the highest is 63.

CONTACTS AND LOCATIONS:
Overall Officials: Özlem Akkoyun Sert, Phd, PT, Study Director — KTO Karatay University; Kamil Yılmaz, Phd, PT, Study Chair — KTO Karatay University; Osman Karaca, MsC,PT, Study Chair — KTO Karatay University; Hasan Gerçek, PT, Study Chair — KTO Karatay University; Bayram Sönmez Ünüvar, MsC, PT, Study Chair — KTO Karatay University; Sinan Bağçacı, Dr, Study Chair — KTO Karatay University; Büşra Alkan, MsC, PT, RA, Study Chair — KTO Karatay University; Melike Akdam, PT, RA, Study Chair — KTO Karatay University; Buse Kılınç, PT, Study Chair — KTO Karatay University
Locations (1):
- KTO Karatay University, Konya, Karatay, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No